CLINICAL TRIAL: NCT02790710
Title: Brief Intervention for OCD Fears
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study has been withdrawn due to reconsideration of study design.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Franklin Schneier, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 7293 (OCD)
Record Dates: First submitted 2016-05-26; First posted 2016-06-06 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Obsessive-compulsive Disorder
Keywords: propanolol; obsessive-compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Propranolol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propanolol (Experimental): Propranolol 40 mg capsule, given once after fear reactivation procedure
  Interventions: Drug: Propanolol
- Placebo capsule (Placebo Comparator): Placebo capsule, given once after fear reactivation procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propanolol — Active treatment
  Other Names: Inderal
  Arms: Propanolol
Drug: Placebo
  Other Names: sugar pill
  Arms: Placebo capsule

SUMMARY:
The study will test the efficacy of propranolol or placebo, administered after reactivation of a previously acquired obsessive-compulsive disorder (OCD) fear, in reducing fear and avoidance in OCD.

DETAILED DESCRIPTION:
Twenty subjects with OCD will be enrolled in the study. Participants will complete baseline assessments of fear and avoidance. Participants will be randomly assigned to a single dose of propranolol 40mg or placebo, administered immediately after a fear reactivation procedure. Primary outcome assessment will be OCD symptoms and avoidance behavior in a behavioral avoidance task 2 weeks after the intervention

ELIGIBILITY:
Inclusion Criteria:

* Principal Diagnosis of Obsessive-Compulsive Disorder

Exclusion Criteria:

* History of other serious psychiatric disorder
* Current Major Depressive Disorder
* Women who are pregnant or nursing
* Current use of psychiatric medication
* Persons planning to start another treatment during the study period
* Any significant medical condition that might increase the risk or participation or use of medications that might negatively interact with propranolol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2023-04 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive-Compulsive Scale | 2 weeks
  Total score on this Clinician-administered measure of OCD symptoms

SECONDARY OUTCOMES:
Behavioral Avoidance Task | 2 weeks
  Total number of steps completed (0-5) on this task assessing avoidance of OCD triggers

CONTACTS AND LOCATIONS:
Overall Officials: Blair Simpson, MD, Study Director — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No